CLINICAL TRIAL: NCT04104126
Title: Blood Flow Restriction Therapy in Achilles Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: s19-01244
Record Dates: First submitted 2019-09-24; First posted 2019-09-26 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Achilles Injuries Tendon
MeSH Terms: interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care Physical Therapy (Active Comparator): Patients with Achilles injury are prescribed PT for their treatment, therefore physical therapy is a standard of care treatment for patients with tendon pathology.
  Interventions: Other: Standard of Care Physical Therapy
- Blood flow restriction (BFR) therapy (Experimental): Blood flow restriction therapy is a blood pressure cuff placed around the desired limb with a handheld device that controls the pressure exerted by the cuff.
  Interventions: Other: Blood flow restriction

INTERVENTIONS:
Other: Standard of Care Physical Therapy — Will receive standard of care physical therapy
  Arms: Standard of Care Physical Therapy
Other: Blood flow restriction — Blood flow restriction therapy is a blood pressure cuff placed around the desired limb with a handheld device that controls the pressure exerted by the cuff. The cuff is placed around the desired limb before a specific exercise, the physical therapist determines the appropriate pressure and time, and the patient completes the exercise as they normally would. The monitor determines the limb occlusion pressure and has an automatic timer that will deflate after the specified time has elapsed.
  Arms: Blood flow restriction (BFR) therapy

SUMMARY:
Blood flow restriction (BFR) therapy is a brief and partial restriction of venous outflow of an extremity during low load resistance exercises. It is a safe and effective method of improving strength in healthy and active individuals, recovering from orthopedic pathologies and procedures. This prospective, randomized study will look at the implications this form of treatment has on the rehabilitation of Achilles injuries.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Achilles Injury
* Must be at least 18 years of age and younger than 65 years of age
* Intention to receive physical therapy as standard of care

Exclusion Criteria:

* Patients with intention to receive standard therapy and not the study therapy
* Patients with impaired circulation, peripheral vascular compromise, previous revascularization of the extremity, or severe hypertension
* Younger than 18 years of age or older than 65
* Legally incompetent or mentally impaired (e.g. minors, Alzheimer's subjects, dementia, etc.)
* Any patient considered a vulnerable subject

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2021-10-08 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
efficacy of blood flow restriction therapy on patients with Achilles injury by measure pre and post blood flow restriction therapy measured by muscle strength | 12 Months
  Measure in increase of strength in the affected leg measured by Biodex.
Measure of pain using Visual Analog Scale (VAS) | 12 Months
  Respondent selects a whole number (0-10 integers) that best reflects the intensity of their pain. For pain intensity, the scale is most commonly anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100 [100-mm scale])

CONTACTS AND LOCATIONS:
Overall Officials: Guillem Gonzalez-Lomas, MD, Principal Investigator — New York Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: Requests should be directed to David.Bloom@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.